CLINICAL TRIAL: NCT06036446
Title: Cervical Cerclage for Short Cervix at 24-26 Weeks of Gestation: a Randomized Controlled Trial
Brief Title: LATe Cerclage in High-risk Pregnancies (LATCH)
Acronym: LATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iRISID-2023-2321
Record Dates: First submitted 2023-08-18; First posted 2023-09-14 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Premature Birth
Keywords: Cervical length; Short cervix; Shortened cervix; Prematurity; Preterm birth; Viability
MeSH Terms: conditions — Premature Birth | interventions — Cerclage, Cervical

STUDY DESIGN:
Intervention Model Description: Randomized trial of cerclage versus no cerclage in singleton high-risk pregnancies with a short TVU CL at 24-26 weeks of gestation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cerclage (Experimental): Cervical cerclage placement with removal during the 36th week of gestation or earlier if clinically indicated.
  Interventions: Procedure: Cervical cerclage; Drug: Vaginal Suppository Progesterone
- Control (Other): Continuing or initiation of vaginal progesterone 200mg daily until 36 weeks of gestation.
  Interventions: Drug: Vaginal Suppository Progesterone

INTERVENTIONS:
Procedure: Cervical cerclage — Transvaginal cervical cerclage placed between 24 0/7 - 26 6/7 weeks of gestation.
  Other Names: Cerclage
  Arms: Cerclage
Drug: Vaginal Suppository Progesterone — Continuing or initiation of vaginal progesterone 200mg daily until 36 weeks of gestation.
  Other Names: Vaginal progesterone

SUMMARY:
The goal of this clinical trial is to determine whether cervical cerclage reduces the risk of preterm birth in patients with a short transvaginal ultrasound (TVU) cervical length (CL) ≤25mm between 24 0/7-26 6/7 weeks.

DETAILED DESCRIPTION:
Singleton high-risk pregnancies < 24 weeks of gestation will be screened for enrollment and randomized, if a short TVU CL (≤25mm) is detected between 24 0/7 - 26 6/7 weeks, to either cervical cerclage or control (no cerclage). Aside from cerclage placement, management of included women will be the same including recommendation for continuing or initiating daily vaginal progesterone 200mg from randomization until 36 6/7 weeks. The primary outcome will be the incidence of preterm birth <37 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old, pregnant, assigned female at birth
* Singleton pregnancy
* TVU CL ≤25mm between 24 0/7 - 26 6/7 weeks of gestation

Exclusion Criteria:

* Initial multifetal gestation with subsequent multifetal pregnancy reduction, or selective fetal termination performed >14 weeks, or cotwin pregnancy loss diagnosed >14 weeks
* Cerclage in situ
* Preterm labor, defined as painful regular uterine contractions and change in cervical dilation
* PPROM
* Active vaginal bleeding
* Suspected intraamniotic infection
* Major fetal structural abnormality or chromosomal disorder
* Placenta previa or accreta
* Other contraindication to cerclage placement
* Participation in another clinical trial related to preterm birth prevention, cerclage, or progesterone

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 329 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of preterm birth <37 weeks | At delivery

SECONDARY OUTCOMES:
Incidence of preterm birth <34 weeks, <32 weeks, and <28 weeks | At delivery
Gestational age at delivery | At delivery
Time interval from randomization to delivery | At delivery
Incidence of preterm prelabor rupture of membranes (PPROM) | At occurrence up to 36 weeks and 6 days of gestation
Incidence of intraamniotic infection | At the time of delivery at any gestational age
  Defined by either presence of clinical criteria (i.e. includes maternal fever [temperature > 100.4 on two occasions at least 30 minutes apart] and one or more of the following: maternal leukocytosis [white blood cell count > 15,000], purulent cervical drainage, or fetal tachycardia), laboratory testing (positive amniotic fluid test result [gram stain, glucose level [<15], or culture results consistent with infection]), or placental pathology demonstrating histologic evidence of placental infection or inflammation.
Neonatal outcomes: incidence of low birthweight (<2500g) | At delivery
Neonatal outcomes: incidence of very low birthweight (<1500g) | At delivery
Neonatal outcomes: incidence of admission to neonatal intensive care unit | At delivery
Neonatal outcomes: composite outcome of incidence of either respiratory distress syndrome, bronchopulmonary dysplasia, grade 3 or 4 intraventricular hemorrhage, necrotizing enterocolitis, culture confirmed sepsis, stillbirth, and neonatal mortality | At least 30 days after delivery, up to 6 months after delivery for outcomes except neonatal mortality

CONTACTS AND LOCATIONS:
Overall Officials: Moti Gulersen, MD, MSc, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Gulersen M, Lenchner E, Nicolaides KH, Otsuki K, Rust OA, Althuisius S, Bornstein E, Berghella V. Cervical cerclage for short cervix at 24 to 26 weeks of gestation: systematic review and meta-analysis of randomized controlled trials using individual patient-level data. Am J Obstet Gynecol MFM. 2023 Jun;5(6):100930. doi: 10.1016/j.ajogmf.2023.100930. Epub 2023 Mar 15. PMID 36924844